CLINICAL TRIAL: NCT03355638
Title: Treatment of Exudative Age-Related Macular Degeneration With Aflibercept Combined With Pranoprofen Eye Drops or Nutraceutical Support With Omega-3: A Randomized Trial
Brief Title: Treatment of CNV With Aflibercept Combined With Pranoprofen Eye Drops or Nutraceutical Support With Omega-3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Andrea Russo, Andrea Russo; MD, PhD, Università degli Studi di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSAIDs_03
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-11

CONDITIONS: Macular Edema
MeSH Terms: conditions — Macular Edema | interventions — aflibercept

STUDY DESIGN:
Intervention Model Description: This was a prospective, randomized, pilot study in 60 patients with treatment-naïve choroidal neovascularization. Patients were randomized 1:1:1 into 3 groups: aflibercept monotherapy, aflibercept plus pranoprofen, or aflibercept plus nutraceutical tablets containing multivitamin antioxidant and mineral supplementation plus omega-3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- aflibercept monotherapy (Active Comparator): All patients received monthly 0.5 mg aflibercept intravitreal injections for 3 months, after which monthly injections were administered pro re nata
  Interventions: Drug: Aflibercept Injection [Eylea]
- aflibercept plus pranoprofen (Experimental): All patients received monthly 0.5 mg aflibercept intravitreal injections for 3 months, after which monthly injections were administered pro re nata. Moreover, patients also self- administered one drop of pranoprofen (Pranoflog; Sifi SpA, Aci Sant'Antonio, CT, Italy) three times a day for 12 months. All patients were followed up for 12 months.
  Interventions: Drug: Aflibercept Injection [Eylea]; Drug: Pranoprofen Eyedrops
- aflibercept plus nutraceutical (Experimental): All patients received monthly 0.5 mg aflibercept intravitreal injections for 3 months, after which monthly injections were administered pro re nata. Moreover, patients were given daily tablets of Omega-3 supplementation (Azyr Mega; Sifi SpA, Aci Sant'Antonio, CT, Italy).
  Interventions: Drug: Aflibercept Injection [Eylea]; Drug: Omega-3 Supplementation

INTERVENTIONS:
Drug: Aflibercept Injection [Eylea] — patients received monthly 0.5 mg aflibercept intravitreal injections for 3 months, after which monthly injections were administered pro re nata
Drug: Pranoprofen Eyedrops — Patients were given a bottle of eyedrops for self-administration of 0.1% pranoprofen (Pranoflog, Sifi SpA, Aci Sant'Antonio, CT, Italy). Pranoprofen dosage was 1 drop in the study eye, 3 times a day, over the 12-month study period
  Arms: aflibercept plus pranoprofen
Drug: Omega-3 Supplementation — Ppatients were given daily tablets of Omega-3 supplementation provided free of charge by the company (Azyr Mega; Sifi SpA, Aci Sant'Antonio, CT, Italy).
  Arms: aflibercept plus nutraceutical

SUMMARY:
To determine whether a combination of intravitreal aflibercept and pranoprofen eyedrops or nutraceutical support provides additional benefit over IVA monotherapy for the treatment of choroidal neovascularization in age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* provision of written informed consent and compliance with study assessments for the full duration of the study
* age > 40 years
* presence of treatment-naïve neovascular AMD.

Exclusion Criteria:

* any previous intravitreal treatment
* previous laser treatment in the study eye
* myopia > 7 diopters in the study eye
* concurrent eye disease in the study eye that could compromise visual acuity (e.g., diabetic retinopathy and advanced glaucoma)
* concurrent corneal epithelial disruption or any condition that would affect the ability of the cornea to heal
* known sensitivity to any component of the formulations being investigated.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Central Retinal Thickness (microns) | 12-month
  Optical Coherence Tomography will be used to assess central retinal thickness.
Visual Acuity (LogMAR) | 12-month
  ETDRS charts will be used to assess best corrected visual acuity

IPD SHARING:
Plan to Share IPD: No